CLINICAL TRIAL: NCT02303015
Title: Toxicity Attributed to Genetic Polymorphisms in Testicular Germ Cell Tumor Survivors
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gedske Daugaard, Professor M.D. DMSc, Rigshospitalet, Denmark
Other Study IDs: DaTeCa01
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Germ Cell Cancer
Keywords: Germ cell cancer; Late toxicity; Renal impairment; Cardiovascular disease
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Renal Insufficiency; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples and /or saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Danish germ cell cancer patients: Danish patients with germ cell cancer diagnosed from 1984 to 2007.

SUMMARY:
The purpose of this study is to identify genetic variations in survivors of testicular cancer and connect these variations to differences in risks of late effects.

DETAILED DESCRIPTION:
Identification of late-effects through questionnaires and linkage to national registries. DNA samples will be gathered through buccal swabs or saliva kits and analysed with whole exome-sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Danish citizen
* Diagnosed with germ cell cancer from 1984 to 2007
* Treated initially at a Danish hospital
* Treated with standard treatment regimens.

Exclusion Criteria:

* Treated initially at a foreign hospital

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Danish patients with germ cell cancer diagnosed 1984-2007.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2014-08; Primary Completion 2023-03 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Renal toxicity (Identify genetic variations predicting renal toxicity) | 1 year
  Identify genetic variations predicting renal toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, MD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of Oncology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No